CLINICAL TRIAL: NCT02802501
Title: Study 200894: A Double-blind, Double-dummy, Randomized, Parallel Group, Placebo-controlled Superiority Study to Evaluate the Efficacy and Safety of Tafenoquine (SB-252263, WR238605) Co-administered With Dihydroartemisinin-piperaquine (DHA-PQP) for the Radical Cure of Plasmodium Vivax Malaria
Brief Title: Efficacy and Safety Study of Tafenoquine (TQ) Co-administered With Dihydroartemisinin-piperaquine (DHA-PQP) for the Radical Cure of Plasmodium Vivax (P. Vivax) Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200894
Record Dates: First submitted 2016-05-26; First posted 2016-06-16 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Malaria, Vivax
Keywords: Safety; Artemisinin Combination Therapy; Efficacy; Tafenoquine; Superiority; Primaquine; Radical cure; Vivax; ACT; Plasmodium vivax malaria; Dihydroartemisinin-piperaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DHA-PQP plus tafenoquine 300 mg single dose (Experimental): Subjects will receive open label DHA-PQP, 3 or 4 tablets per day (according to the body weight) from Day 1 to Day 3. They will receive double-blind 300 mg single dose of tafenoquine (TQ) on Day 1 and matched-placebo for primaquine (PQ) from Day 1 to Day 14.
  Interventions: Drug: Tafenoquine; Drug: Matched-Placebo for Primaquine; Drug: Dihydroartemisinin-piperaquine (DHA-PQP); Drug: ACT plus PQ (Rescue medication); Drug: PQ (End of study treatment)
- DHA-PQP plus primaquine 15 mg for 14 days (Active Comparator): Subjects will receive open label DHA-PQP, 3 or 4 tablets per day (according to body weight) from Day 1 to Day 3. They will receive double-blind 15 mg primaquine (PQ) from Day 1 to Day 14 and matched-placebo for tafenoquine (TQ) on Day 1.
  Interventions: Drug: Matched-Placebo for Tafenoquine; Drug: Primaquine; Drug: Dihydroartemisinin-piperaquine (DHA-PQP); Drug: ACT plus PQ (Rescue medication); Drug: PQ (End of study treatment)
- DHA-PQP alone (placebo arm) (Placebo Comparator): Subjects will receive open label DHA-PQP, 3 or 4 tablets per day (according to body weight) from Day 1 to Day 3. They will receive double-blind matched-placebo for tafenoquine (TQ) on Day 1 and matched-placebo for primaquine (PQ) from Day 1 to Day 14.
  Interventions: Drug: Matched-Placebo for Tafenoquine; Drug: Matched-Placebo for Primaquine; Drug: Dihydroartemisinin-piperaquine (DHA-PQP); Drug: ACT plus PQ (Rescue medication); Drug: PQ (End of study treatment)

INTERVENTIONS:
Drug: Tafenoquine — This intervention is provided as tablet containing 150 mg of tafenoquine. Two tablets of this formulation will be administered orally with water as a single dose after a meal. Dose will be taken at least 3 hours after DHA-PQP.
  Arms: DHA-PQP plus tafenoquine 300 mg single dose
Drug: Matched-Placebo for Tafenoquine — This intervention contains tafenoquine matched-placebo. Two tablets of this formulation will be administered orally with water as a single dose after a meal. Dose will be taken at least 3 hours after DHA-PQP.
  Arms: DHA-PQP alone (placebo arm); DHA-PQP plus primaquine 15 mg for 14 days
Drug: Primaquine — This intervention is provided as over-encapsulated tablet containing 15 mg of primaquine. One capsule of this formulation will be administered orally with water as a single dose after a meal for 14 days. Dose will be taken at least 3 hours after DHA-PQP (Days 1, 2 and 3).
  Arms: DHA-PQP plus primaquine 15 mg for 14 days
Drug: Matched-Placebo for Primaquine — This intervention contains primaquine matched-placebo. One capsule of this formulation will be administered orally with water as a single dose after a meal for 14 days. Dose will be taken at least 3 hours after DHA-PQP (Days 1, 2 and 3).
  Arms: DHA-PQP alone (placebo arm); DHA-PQP plus tafenoquine 300 mg single dose
Drug: Dihydroartemisinin-piperaquine (DHA-PQP) — This formulation is provided as tablet containing 320 mg of piperaquine tetrasphosphate (as the tetrahydrate; PQP) and 40 mg dihydroartemisinin (DHA). This tablet will be administered orally as single dose for 3 days. For subjects weighing <75 kg, 3 tablets will be administered per day. For subjects weighing >=75 kg, 4 tablets will be administered per day. Dose will be taken at least 3 hours after last food intake. No food will be allowed for at least 3 hours after dosing.
Drug: ACT plus PQ (Rescue medication) — Subjects with relapse during the 180 day follow up period will be given an ACT plus PQ 0.5 mg/kg for 14 days as rescue medication.
Drug: PQ (End of study treatment) — Subjects who do not relapse during the study will receive PQ 0.5mg/kg for 14 days at the end of the study.

SUMMARY:
Tafenoquine (TQ) is an 8-aminoquinoline anti-malarial drug which is in development as a single-dose treatment for the radical cure of P.vivax malaria when given with standard doses of chloroquine. Currently, the only available drug for radical cure is primaquine (PQ) which requires administration over 14 days, resulting in poor compliance. In Indonesia, chloroquine has been replaced by artemisinin-based combination therapy (i.e. ACTs) due to widespread chloroquine resistance. This study will evaluate the efficacy and safety of a single dose of tafenoquine when co-administered with an ACT (i.e. DHA-PQP). This single-center, double-blind, double-dummy, randomized study will test the superiority of DHA-PQP plus TQ against DHA-PQP alone in the prevention of P. vivax malaria relapse at 6 months. The study will be conducted in male Indonesian soldiers diagnosed with P.vivax malaria on return from deployment to a malarious region of Indonesia. A PQ plus DHA-PQP comparator arm is included to provide an informal comparison against the standard 14 day treatment for P.vivax malaria in Indonesia. Subjects who are glucose-6-phosphate dehydrogenase deficient (G6PD deficient) will be excluded due to the risk of acute hemolysis following dosing with 8-aminoquinolines drugs. Subjects who have a recurrence of P.vivax malaria during the study will be treated with an ACT plus PQ (0.5mg/kg for 14 days), in line with local treatment guidelines. At the end of the 6 month follow up period, any subject who has not relapsed will be given open label PQ (0.5mg/kg daily for 14 days) to minimize the likelihood of relapse after the study. Approximately 200 subjects will be screened to achieve 150 randomized subjects. The total duration of study for each subject will be 180-195 days. This study is being carried out to support registration of TQ in Indonesia and other countries where ACTs are first line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects >=18 years at the time of signing the informed consent.
* The subject has a positive Giemsa smear for P. vivax (mixed infection with P.falciparum is acceptable).
* The subject has a parasite density of >20 per microliter.
* Glucose-6-phosphate dehydrogenase (G6PD) normal using a suitable qualitative assessment, for example, nicotinamide adenine dinucleotide phosphate (NADPH) qualitative fluorescent spot test (Trinity Biologicals, United States of America).
* The subject has a QTcF of <450 millisecond (msec). Note: Reading based on an average of triplicate ECGs obtained over a brief recording period by machine.
* The subject is willing and able to comply with the study protocol.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* Severe P.vivax malaria as defined by World Health Organization (WHO) criteria.
* Severe vomiting (no food or inability to take food during the previous 8 hours).
* Screening hemoglobin (Hb) concentration <8 grams per deciliter.
* Liver function test ALT >2 times upper limit of Normal (ULN).
* Any clinically significant concurrent illness (for example, pneumonia, septicemia), significant pre-existing conditions (for example, renal disease, malignancy, Type 1 diabetes), conditions that may affect absorption of study treatment (for example, vomiting, severe diarrhea), or clinical signs and symptoms of severe cardiovascular disease (for example, uncontrolled congestive heart failure, severe coronary artery disease).
* History of hypersensitivity, allergy or adverse reactions to Dihydroartemisinin (DHA) or other artemisinins, piperaquine, tafenoquine or primaquine.
* Subject has previously received treatment with tafenoquine, or has received treatment with any other investigational drug within 30 days of study entry or within 5 half-lives, whichever is longer.
* Subject has taken anti-malarials (for example, ACTs, mefloquine, primaquine, quinacrine) or drugs with anti-malarial activity within the past 30 days.
* Subjects who will likely require the use of medications from the prohibited medications list or have taken them in the past 30 days which include the following medications and medication classes: Drugs with hemolytic potential, Drugs known to prolong the QT corrected (QTc) interval including: Antiarrhythmics; Neuroleptics and antidepressive agents; Certain antimicrobial agents, including agents of the following classes: macrolides, fluroquinolones imidazole and triazole antifungal agents and also pentamidine and saquinavir; Certain non-sedating antihistamines; Cisapride, droperidol, domperidone, bepridil, diphemanil, probucol, levomethadyl, methadone, vinca alkaloids, arsenic trioxide.
* The biguanides: phenformin and buformin (but excluding metformin).
* Drugs that are substrates of the renal transporters organic cation transporter 2 (OCT2), multidrug and toxin extrusion protein 2 (MATE1) and multidrug and toxin extrusion protein 2 (MATE2) and have a narrow therapeutic index (for example, the antiarrhythmic agents: dofetilide, procainamide and pilsicainide).
* Anticipated to be unable to consume daily study treatment under direct supervision by the research team.
* Previous participation in the present clinical trial, that is, subjects experiencing relapse during or after the study period may not be enrolled as a new subject.
* History of illicit drug abuse or heavy alcohol intake, such that full participation in the study could be compromised.
* Any contraindication in the opinion of the Investigator to DHA-PQP or primaquine administration such as: Family history of sudden unexplained death (DHA-PQP); Known congenital QT corrected (QTc) prolongation (DHA-PQP); Known history of a medical condition known to prolong the QT interval: for example, myxoedema, cardiomyopathies, recent myocardial infarction (DHA-PQP); History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia (DHA-PQP); Cardiac illnesses predisposing to arrhythmias for example, severe hypertension, left ventricular hypertrophy, cardiomyopathies, cardiac failure with reduced ejection fraction (DHA-PQP); Presence of an electrolyte disturbance particularly hypokalemia, hypocalcemia, hypomagnesemia (DHA-PQP); Rheumatoid arthritis, lupus erythematosus and other systemic conditions that may cause granulocytopenia (primaquine); History of hemolytic anemia, methemoglobinemia and leucopenia (primaquine).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sutanto I, Soebandrio A, Ekawati LL, Chand K, Noviyanti R, Satyagraha AW, Subekti D, Santy YW, Crenna-Darusallam C, Instiaty I, Budiman W, Prasetya CB, Lardo S, Elyazar I, Duparc S, Cedar E, Rolfe K, Fernando D, Berni A, Jones S, Kleim JP, Fletcher K, Sharma H, Martin A, Taylor M, Goyal N, Green JA, Tan LK, Baird JK. Tafenoquine co-administered with dihydroartemisinin-piperaquine for the radical cure of Plasmodium vivax malaria (INSPECTOR): a randomised, placebo-controlled, efficacy and safety study. Lancet Infect Dis. 2023 Oct;23(10):1153-1163. doi: 10.1016/S1473-3099(23)00213-X. Epub 2023 May 23. PMID 37236221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single center randomized, double-blind, parallel group study to evaluate the efficacy and safety of tafenoquine co-administered with DHA-PQP for the radical cure of P.vivax malaria in Indonesian soldiers. Participants with microscopy-confirmed P.vivax were recruited at 2malaria-free bases in Java following deployment to Indonesian Papua.
Pre-assignment Details: A total of 164 participants were screened of whom 14 failed during screening and 150 were randomized to receive dihydroartemisinin-piperaquine (DHA-PQP) only, tafenoquine+DHA-PQP and primaquine+DHA-PQP in a ratio of 1:1:1.
Groups:
- DHA-PQP Only: Participants received either 3 tablets (body weight: <75 kilograms [kg]) or 4 tablets (body weight: >=75 kg) per day of open-label DHA-PQP on Days 1 to 3. Participants also received blinded treatment with tafenoquine matched placebo tablet administered as a single oral dose and once daily oral doses of primaquine matched placebo for 14 days. Blinded treatment started on Day 1 or Day 2. Participants who did not relapse before Day 180 were administered 0.5 milligrams (mg)/kg open-label primaquine once daily for 14 days after completion of the double-blind phase.
- Tafenoquine+ DHA-PQP: Participants received either 3 tablets (body weight: <75 kg) or 4 tablets (body weight: >=75 kg) per day of open-label DHA-PQP on Days 1 to 3. Participants also received blinded treatment with tafenoquine 300 mg administered as a single oral dose and once daily oral doses of primaquine matched placebo for 14 days. Blinded treatment started on Day 1 or 2. Participants who did not relapse before Day 180 were administered 0.5 mg/kg open-label primaquine once daily for 14 days after completion of the double-blind phase.
- Primaquine+DHA-PQP: Participants received either 3 tablets (body weight: <75 kg) or 4 tablets (body weight: >=75 kg) per day of open-label DHA-PQP on Days 1 to 3. Participants also received blinded treatment with tafenoquine matched placebo administered as a single oral dose and once daily oral doses of primaquine 15 mg for 14 days. Participants who did not relapse before Day 180 were administered 0.5 mg/kg open-label primaquine once daily for 14 days after completion of the double-blind phase.
Period: Double-blind (Up to Day 180)
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0
Period: Open-Label (Day 180 to Day 195)
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Started | 6 (Participants who had no relapse prior to Day 180 received open-label Primaquine) | 12 (Participants who had no relapse prior to Day 180 received open-label Primaquine) | 26 (Participants who had no relapse prior to Day 180 received open-label Primaquine)
Completed | 6 | 12 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.3 (4.34) | 29.4 (5.10) | 28.6 (5.56) | 28.8 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 50 | 50 | 50 | 150
Race/Ethnicity, Customized [Number; unit: Participants]
  ASIAN - SOUTH EAST ASIAN HERITAGE | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Relapse-free Efficacy at Six Months After Administration of Tafenoquine With DHA-PQP and DHA-PQP Alone
Description: A participant was considered to have demonstrated relapse-free efficacy at 6 months if: a) Participant had non-zero Plasmodium vivax (P.vivax) asexual parasite count at Baseline (Day 1), b) Participant demonstrated initial clearance of P.vivax parasitemia, c) Participant had no positive asexual P.vivax parasite count at any assessment prior to or on study Day 180 following initial parasite clearance, d) Participants did not take a concomitant medication with anti-malarial activity (excluding study treatment) at any point between Study Day 1 and their last parasite assessment, e) Participant was parasite-free at 6 months. The percentage of participants who were relapse-free at 6 months post dose has been presented.
Time Frame: 6 months post-dose
Population: Microbiologic Intent-to-Treat (mITT) Population consisted of all randomized participants who received at least one dose of blinded study treatment and had microscopically confirmed P. vivax parasitamia at Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP
Number analyzed (Participants) | 50 | 50
Percentage of participants | 12 | 22
Statistical Analysis 1: Comparison: DHA-PQP Only vs Tafenoquine+ DHA-PQP; Test type: Superiority; p < 0.001, Cox Proportional Hazard; Hazard Ratio (HR) = 0.444, 95% CI 2-sided [0.285 to 0.693] — If hazard ratio was found to be <1 then there are lower chances of relapse with Tafenoquine+DHA-PQP compared to DHA-PQP only

2. Secondary Outcome: Percentage of Participants With Relapse-free Efficacy at Six Months After Administration of Tafenoquine With DHA-PQP and Primaquine+DHA-PQP
Description: A participant was considered to have demonstrated relapse-free efficacy at 6 months if: a) Participant had non-zero P. vivax asexual parasite count at Baseline (Day 1), b) Participant demonstrated initial clearance of P.vivax parasitemia, c) Participant had no positive asexual P.vivax parasite count at any assessment prior to or on study Day 180 following initial parasite clearance, d) Participants did not take a concomitant medication with anti-malarial activity (excluding study treatment) at any point between Study Day 1 and their last parasite assessment, e) Participant was parasite-free at 6 months. The percentage of participants who were relapse-free at 6 months post dose has been presented.
Time Frame: 6 months post-dose
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50
Percentage of participants | 22 | 52
Statistical Analysis 1: Comparison: Tafenoquine+ DHA-PQP vs Primaquine+DHA-PQP; Test type: Superiority; Hazard Ratio (HR) = 1.722, 95% CI 2-sided [1.031 to 2.875] — If hazard ratio was found to be >1 then there are higher chances of relapse with Tafenoquine+DHA-PQP compared to Primaquine+DHA-PQP

3. Secondary Outcome: Percentage of Participants With Relapse-free Efficacy at Six Months After Administration of Primaquine With DHA-PQP and DHA-PQP Alone
Description: as for outcome 2
Time Frame: 6 months post-dose
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | DHA-PQP Only | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50
Percentage of participants | 12 | 52
Statistical Analysis 1: Comparison: DHA-PQP Only vs Primaquine+DHA-PQP; Test type: Superiority; Hazard Ratio (HR) = 0.258, 95% CI 2-sided [0.155 to 0.431] — If hazard ratio was found to be <1 then there are lower chances of relapse with Primaquine+DHA-PQP compared to DHA-PQP only

4. Secondary Outcome: Percentage of Participants With Relapse-free Efficacy at Four Months After Administration of Tafenoquine With DHA-PQP and DHA-PQP Alone
Description: A participant was considered to have demonstrated recurrence-free efficacy at 4 months if: a) Participant had non-zero P. vivax asexual parasite count at Baseline, b) Participant demonstrated initial clearance of P.vivax parasitemia, c) Participant had no positive asexual P.vivax parasite count at any assessment prior to or on Study Day 135 following initial parasite clearance, d) Participants did not take a concomitant medication with anti-malarial activity (excluding study treatment) at any point between Study Day 1 and their first parasite assessment after Study Day 105 (up to and including Study Day 135), e) Participant was parasite-free at 4 months. The rate of relapse-free efficacy was estimated by Kaplan-Meier methodology. The percentage of participants who were relapse-free at 4 months post dose has been presented.
Time Frame: 4 months post-dose
Population: mITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP
Number analyzed (Participants) | 50 | 50
Percentage of participants | 16 | 28
Statistical Analysis 1: Comparison: DHA-PQP Only vs Tafenoquine+ DHA-PQP; Test type: Superiority; Hazard Ratio (HR) = 0.433, 95% CI 2-sided [0.273 to 0.686] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to Relapse of P. Vivax Malaria
Description: Relapse is defined by a positive blood smear with or without vivax symptoms. Relapse is described as any recurrence of P. vivax malaria after clearance of the initial infection. The time to relapse (number of days between the date of first positive count and date of Study Day 1) was analyzed by the Kaplan-Meier method. The median number of days to relapse along with 95 percent (%) confidence interval (CI) has been presented for each treatment group.
Time Frame: Up to Day 180
Population: mITT Population.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Days | 81.5 [74.0 to 88.0] | 96.0 [88.0 to 117.0] | NA [90.0 to NA] — NA indicates median and 95% CI (upper limit) could not be derived, as <50% of participants experienced the event within the treatment arm.

6. Secondary Outcome: Time to Fever Clearance
Description: Time to fever clearance is defined as time from first dose of treatment to the time when body temperature falls to normal and remains normal for at least 48 hours up to the Day 7 visit. Fever clearance is considered to have been achieved once an initial temperature of greater than 37.4 degree Celsius is reduced to a value less than or equal to 37.4 degree Celsius, in the absence of value greater than 37.4 degree Celsius in the following 48 hours up to Day 7 visit. The time taken to achieve fever clearance was analyzed by Kaplan-Meier method.
Time Frame: Up to Day 7
Population: mITT Population.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Hours | 16.5 [14.1 to 17.3] | 15.8 [13.1 to 18.8] | 16.8 [14.6 to 17.8]

7. Secondary Outcome: Time to Parasite Clearance
Description: Parasite clearance time is defined as time needed to clear asexual parasite from the blood that is, parasite numbers falling below the limit of detection in the thick blood smear and remaining undetectable after >= 6 hours later. The time to achieve parasite clearance was analyzed by Kaplan-Meier method.
Time Frame: Up to Day 8
Population: mITT Population.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Hours | 18.1 [18.0 to 18.7] | 18.1 [18.0 to 18.3] | 18.0 [18.0 to 18.1]

8. Secondary Outcome: Number of Participants With Recrudescence
Description: Recrudescence was defined as blood stage treatment failure. A participant was considered to have had a recrudescence if both of the following were true: 1) if participant had a positive P. vivax asexual parasite count at Baseline and demonstrated clearance (i.e. two negative asexual P. vivax parasite counts, with at least 6 hours between the counts, and no positive counts in the interval); 2) Participant had a positive genetically homologous asexual P. vivax parasite count on or before Study Day 14, after their zero count in days 1 to 5.
Time Frame: Up to Day 14
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Double-blind Treatment Phase
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function, other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 180
Population: Safety Population consisted of all randomized participants who received at least one dose of blinded study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Any AEs | 41 | 41 | 34
  Any SAEs | 1 | 2 | 2

10. Secondary Outcome: Number of Participants With Chemistry Values Outside Clinical Concern Range
Description: Blood samples were collected at indicated time points to analyze following chemistry parameters: alanine aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Bilirubin, Creatine Kinase, Creatinine, Indirect Bilirubin and Urea. Clinical concern range for the parameters included ALT and AST (high: >3 times Upper Limit of Normal [ULN]), ALP (high: >2.5 times ULN), bilirubin and indirect bilirubin (high: >1.5 times ULN), creatine kinase (high: >5 times ULN), creatinine (high: >3 times ULN) and urea (high: >11.067 millimoles per Liter [mmol/L]. Data for any time on treatment has been presented.
Time Frame: Up to Day 120
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  ALT, High | 1 | 3 | 0
  ALP, High | 1 | 0 | 0
  AST, High | 0 | 1 | 0
  Bilirubin, High | 4 | 6 | 4
  Creatine Kinase, High | 7 | 6 | 6
  Creatinine, High | 0 | 0 | 0
  Indirect bilirubin, High | 1 | 1 | 1
  Urea, High | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Hematology Values Outside Clinical Concern Range
Description: Blood samples were collected to analyze the following hematology parameters: Hemoglobin, lymphocytes and Platelet count. The clinical concern ranges for the parameters included: hemoglobin (low: <7 grams per deciliter), lymphocytes: (low: <0.5x10^9 cells per liter and high: >4x10^9 cells per liter),and platelets (low: <50x10^9 cells per liter). Data for any time on treatment has been presented.
Time Frame: Up to Day 120
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Hemoglobin, Low | 0 | 0 | 0
  Lymphocytes, High | 3 | 4 | 2
  Lymphocytes, Low | 0 | 0 | 1
  Platelets, Low | 0 | 1 | 0

12. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Values Outside Clinical Concern Range-QT Interval Corrected Using Fredericia's Formula (QTcF)
Description: 12-lead ECG was obtained at indicated time points using an automated ECG machine that measured QTcF. Clinical concern range included:absolute QTcF interval (upper: >480 milliseconds) and increase from Baseline in QTcF (upper: >=60 milliseconds). Data for maximum post-Baseline increase >=60 and >480 milliseconds has been presented.
Time Frame: Up to Day 28
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants | 2 | 3 | 1

13. Secondary Outcome: Change From Baseline in QT Interval Corrected by Fridericia's Formula (QTcF)
Description: 12-lead ECG was obtained at indicated time points using an automated ECG machine that measured QTcF interval. Change from Baseline is calculated as Post-Dose Visit Value minus Baseline value. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1), Day 3: 4 hours post DHA-PQP dose, Days 7 and 28
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Milliseconds
  Day 3: 4 hours post DHA-PQP dose | 35.3 (24.81) | 44.5 (22.96) | 40.8 (17.22)
  Day 7 | 11.5 (14.95) | 12.2 (13.97) | 16.5 (16.67)
  Day 28 | 2.4 (15.00) | 7.5 (13.70) | 10.2 (14.41)

14. Secondary Outcome: Number of Participants With Worst Case Body Temperature Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Body temperature was measured with participants in semi-supine position after 5 minutes of rest. Data was categorized as: body temperature 'low: <36.5 degrees celsius', 'high: >37.3 degrees celsius' and 'To Normal or No change'. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose vital sign value category was unchanged (e.g.,High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1) and up to Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  To Low | 42 | 38 | 42
  To Normal or No change | 3 | 7 | 5
  To High | 10 | 14 | 6

15. Secondary Outcome: Number of Participants With Worst Case Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: SBP and DBP were measured with participants in semi-supine position after 5 minutes of rest. Data was categorized as: systolic blood pressure (SBP) (low: <90 and high: >120 millimeters of mercury [mmHg]); diastolic blood pressure (DBP) (low: <60 and high: >80 mmHg); and 'To Normal or No change'. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose vital sign value category was unchanged (e.g.,High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1) and up to Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  SBP, To Low | 0 | 1 | 0
  SBP, To Normal or No change | 19 | 21 | 25
  SBP, To High | 31 | 29 | 25
  DBP, To Low | 11 | 9 | 15
  DBP, To Normal or No change | 16 | 20 | 16
  DBP, To High | 28 | 25 | 28

16. Secondary Outcome: Number of Participants With Worst Case Pulse Rate Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Pulse rate was measured with participants in semi-supine position after 5 minutes of rest. Data was categorized as: pulse rate low: <60 beats per minute [bpm], high: >100 bpm and 'To normal or No change'. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose vital sign value category was unchanged (e.g.,High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1) and up to Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  To Low | 19 | 26 | 23
  To Normal or No change | 25 | 23 | 26
  To High | 7 | 6 | 3

17. Secondary Outcome: Number of Participants With Worst Case Respiratory Rate Results Relative to Normal Range Post-Baseline Relative to Baseline
Description: Respiratory rate was measured with participants in semi-supine position after 5 minutes of rest. Data was categorized as: respiratory rate low: <12 breaths per minute', high: >18 breaths per minute and 'To normal or No change'. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there was no change in their category. Participants whose vital sign value category was unchanged (e.g.,High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%.Day 1 was considered as Baseline. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1) and up to Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  To Low | 0 | 0 | 0
  To Normal or No change | 41 | 41 | 40
  To High | 9 | 9 | 10

18. Secondary Outcome: Number of Participants With Gastrointestinal AEs
Description: The number of participants with gastrointestinal AEs: nausea, vomiting, diarrhea, dyspepsia, abdominal distension, abdominal discomfort and constipation has been presented.
Time Frame: Up to Day 180
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Nausea | 5 | 4 | 3
  Vomiting | 6 | 5 | 1
  Diarrhea | 5 | 2 | 2
  Dyspepsia | 2 | 3 | 4
  Abdominal distension | 1 | 1 | 1
  Abdominal discomfort | 0 | 0 | 2
  Constipation | 0 | 1 | 0

19. Secondary Outcome: Change From Baseline in Methemoglobin/ Total Hemoglobin
Description: Blood samples were collected for the assessment of methemoglobin/Total Hemoglobin (Hb). Methemoglobin is a type of Hb in the form of metalloprotein that cannot bind with oxygen, measured as percentage of methemoglobin in total hemoglobin. Change from Baseline is calculated as Post-Dose Visit Value minus Baseline value. Day 1 was considered as Baseline.
Time Frame: Baseline (Day 1) and Days 2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,18,20,21,22,24,26,28 and 60
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Percentage of Methemoglobin in total Hb
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 48 | 50 | 50
Percentage of Methemoglobin in total Hb
  Day 2, n=48, 50, 50 | -0.13 (0.234) | -0.07 (0.341) | -0.06 (0.260)
  Day 3, n=48, 50, 50 | -0.16 (0.211) | -0.04 (0.323) | 0.01 (0.270)
  Day 4, n=48, 50, 50 | -0.16 (0.228) | 0.06 (0.367) | 0.28 (0.438)
  Day 5, n=48, 50, 50 | -0.18 (0.244) | 0.12 (0.382) | 0.62 (0.714)
  Day 6, n=46, 49, 50: number analyzed (Participants) | 46 | 49 | 50
  Day 6, n=46, 49, 50 | -0.15 (0.204) | 0.16 (0.437) | 0.91 (0.869)
  Day 7, n=48, 50, 50 | -0.19 (0.248) | 0.19 (0.454) | 1.20 (1.213)
  Day 8, n=46, 48, 48: number analyzed (Participants) | 46 | 48 | 48
  Day 8, n=46, 48, 48 | -0.12 (0.224) | 0.23 (0.487) | 1.41 (1.329)
  Day 9, n=46, 47, 47: number analyzed (Participants) | 46 | 47 | 47
  Day 9, n=46, 47, 47 | -0.13 (0.245) | 0.24 (0.426) | 1.53 (1.325)
  Day 10, n=47, 45, 49: number analyzed (Participants) | 47 | 45 | 49
  Day 10, n=47, 45, 49 | -0.16 (0.279) | 0.24 (0.456) | 1.69 (1.314)
  Day 11, n=47, 44, 49: number analyzed (Participants) | 47 | 44 | 49
  Day 11, n=47, 44, 49 | -0.13 (0.232) | 0.18 (0.445) | 1.82 (1.324)
  Day 12, n=47, 47, 50: number analyzed (Participants) | 47 | 47 | 50
  Day 12, n=47, 47, 50 | -0.13 (0.256) | 0.18 (0.404) | 1.92 (1.436)
  Day 13, n=48, 48, 48: number analyzed (Participants) | 48 | 48 | 48
  Day 13, n=48, 48, 48 | -0.14 (0.256) | 0.18 (0.419) | 2.02 (1.409)
  Day 14, n=48, 50, 50 | -0.18 (0.243) | 0.12 (0.404) | 2.01 (1.436)
  Day 15, n=17, 22, 14: number analyzed (Participants) | 17 | 22 | 14
  Day 15, n=17, 22, 14 | -0.08 (0.213) | 0.00 (0.363) | 2.13 (1.019)
  Day 16, n=43, 48, 47: number analyzed (Participants) | 43 | 48 | 47
  Day 16, n=43, 48, 47 | -0.12 (0.216) | 0.12 (0.369) | 1.84 (1.259)
  Day 18, n=46, 48, 49: number analyzed (Participants) | 46 | 48 | 49
  Day 18, n=46, 48, 49 | -0.12 (0.246) | 0.11 (0.357) | 1.29 (0.982)
  Day 20, n=42, 49, 48: number analyzed (Participants) | 42 | 49 | 48
  Day 20, n=42, 49, 48 | -0.09 (0.260) | 0.06 (0.362) | 0.80 (0.744)
  Day 21, n=43, 48, 48: number analyzed (Participants) | 43 | 48 | 48
  Day 21, n=43, 48, 48 | -0.07 (0.382) | 0.03 (0.262) | 0.69 (0.680)
  Day 22, n=45, 49, 48: number analyzed (Participants) | 45 | 49 | 48
  Day 22, n=45, 49, 48 | -0.13 (0.294) | 0.01 (0.293) | 0.49 (0.565)
  Day 24, n=41, 46, 47: number analyzed (Participants) | 41 | 46 | 47
  Day 24, n=41, 46, 47 | -0.11 (0.258) | 0.03 (0.329) | 0.41 (0.424)
  Day 26, n=44, 45, 47: number analyzed (Participants) | 44 | 45 | 47
  Day 26, n=44, 45, 47 | -0.17 (0.256) | 0.03 (0.279) | 0.19 (0.347)
  Day 28, n=47, 50, 50: number analyzed (Participants) | 47 | 50 | 50
  Day 28, n=47, 50, 50 | -0.15 (0.248) | 0.01 (0.284) | 0.08 (0.314)
  Day 60, n=47, 50, 49: number analyzed (Participants) | 47 | 50 | 49
  Day 60, n=47, 50, 49 | -0.11 (0.260) | -0.07 (0.326) | -0.01 (0.245)

20. Secondary Outcome: Number of Participants With Protocol-defined SAE (Hemoglobin Drop)
Description: Blood samples were collected at indicated time points to analyze the hemoglobin level. Hemoglobin drop is defined as any one of the following occurring in the first 15 days of the study: a relative hemoglobin decrease of >=30% from Baseline, or an absolute hemoglobin decrease of >3 grams per liter from Baseline, or a drop in absolute hemoglobin to <7.0 grams per decilter (g/dL). Number of participants with a protocol-defined hemoglobin SAEs has been presented.
Time Frame: Days 3, 5, 7, and 14
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Day 3 | 0 | 0 | 0
  Day 5 | 0 | 0 | 0
  Day 7 | 0 | 0 | 0
  Day 14 | 0 | 0 | 0

21. Secondary Outcome: Oral Clearance (CL/F) of Tafenoquine When Co-administered With DHA-PQP
Description: Blood samples were collected at the indicated time points for the determination of oral clearance following tefenoquine co-administered with DHA-PQP and was to be calculated by covariate analysis.
Time Frame: Up to Day 60
Reporting Status: Not Posted, anticipated posting 2021-05

22. Secondary Outcome: Volume of Distribution (V/F) of Tafenoquine When Co-administered With DHA-PQP
Description: Blood samples were collected at the indicated time points for the determination of volume of distribution following tefenoquine co-administered with DHA-PQP and was to be calculated by covariate analysis.
Time Frame: Up to Day 60
Reporting Status: Not Posted, anticipated posting 2021-05

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the study treatment up to Day 180 for double-blind treatment phase and from Day 180 to Day 195 for open-label treatment phase
Description: AEs and SAEs were collected in the Safety Population for a) Open Label DHA-PQP phase, b) Double-blind treatment phase and c) Open-label phase comprised of participants who did not relapse during the double-blind phase and went onto the open-label primaquine phase.
Groups:
- DHA-PQP Only (Open-label Primaquine Phase); Tafenoquine 300 mg+DHA-PQP (Open-label Primaquine Phase): Participants received either 3 tablets (body weight: <75 kg) or 4 tablets (body weight: >=75 kg) per day of open-label DHA-PQP on Days 1 to 3. Participants also received oral doses of primaquine matched placebo once daily for 14 days. Participants who did not relapse before Day 180 were administered 0.5 mg/kg open-label primaquine once daily for 14 days after completion of the double-blind phase.
- Primaquine 15 mg+DHA-PQP (Open-label Primaquine Phase): Participants received either 3 tablets (body weight: <75 kg) or 4 tablets (body weight: >=75 kg) per day of open-label DHA-PQP on Days 1 to 3. Participants also received oral doses of primaquine 15 mg once daily for 14 days. Participants who did not relapse before Day 180 were administered 0.5 mg/kg open-label primaquine once daily for 14 days after completion of the double-blind phase.
Arm/Group | DHA-PQP Only | Tafenoquine+ DHA-PQP | Primaquine+DHA-PQP | DHA-PQP Only (Open-label Primaquine Phase) | Tafenoquine 300 mg+DHA-PQP (Open-label Primaquine Phase) | Primaquine 15 mg+DHA-PQP (Open-label Primaquine Phase)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/6 | 0/12 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/50 | 2/50 | 0/6 | 1/12 | 0/26
Other Adverse Events (participants affected / at risk) | 32/50 | 36/50 | 27/50 | 0/6 | 1/12 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DHA-PQP Only (N=50) | Tafenoquine+ DHA-PQP (N=50) | Primaquine+DHA-PQP (N=50) | DHA-PQP Only (Open-label Primaquine Phase) (N=6) | Tafenoquine 300 mg+DHA-PQP (Open-label Primaquine Phase) (N=12) | Primaquine 15 mg+DHA-PQP (Open-label Primaquine Phase) (N=26)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DHA-PQP Only (N=50) | Tafenoquine+ DHA-PQP (N=50) | Primaquine+DHA-PQP (N=50) | DHA-PQP Only (Open-label Primaquine Phase) (N=6) | Tafenoquine 300 mg+DHA-PQP (Open-label Primaquine Phase) (N=12) | Primaquine 15 mg+DHA-PQP (Open-label Primaquine Phase) (N=26)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 11 (13) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (7) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (9) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 4 (4) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT02802501/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT02802501/SAP_001.pdf